CLINICAL TRIAL: NCT06365502
Title: A Multicenter, Prospective, Open-label, Controlled, Randomized Trial of Preventive Drug-coated Balloon Angioplasty in Vulnerable Atherosclerotic Plaque (RESTORE Trial)
Brief Title: Preventive Drug-coated Balloon Angioplasty in Vulnerable Atherosclerotic Plaque (RESTORE Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Yu Bo, Director, Cardiology Department, the 2nd Affiliated Hospital of Harbin Medical University, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-156
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB treatment (Experimental): Non-flow limited vulnerable plaque will be treated by drug-coated balloon when the enrolled individual is randomized into DCB treatment group. The individual located in DCB treatment will receive guideline-directed medical treatment.
  Interventions: Device: Drug-coated balloon; Drug: Guideline-directed medical treatment
- Guideline-directed medical treatment (Active Comparator): Non-flow limited vulnerable plaque will be left with no intervention when the individual is randomized into guideline-directed medical treatment group. The individual will receive guideline-directed medical treatment alone.
  Interventions: Drug: Guideline-directed medical treatment

INTERVENTIONS:
Device: Drug-coated balloon — Non-culprit lesion will be pretreated before DCB treatment. The bail-out stent treatment is permitted if pretreatment failed.
  Arms: DCB treatment
Drug: Guideline-directed medical treatment — All individuals will receive guideline-directed medical treatment.

SUMMARY:
The objective of this multicenter, prospective, open-label, controlled, randomized trial is to demonstrate the superiority of drug-coated balloon (DCB) treatment on non-flow limited vulnerable plaque as compared to guideline-directed medical therapy (GDMT) in improving clinical cardiovascular outcomes in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 80 years of age
2. Subject must present with acute myocardial infarction or unstable angina planned for PCI
3. Successful stent implantation (i.e., residual stenosis less than 20%) must be done in culprit lesions and any lesions with ischemia evidence (e.g., QFR equal or less than 0.8)
4. Subject must have at least one native non-culprit lesion with visually estimated stenosis of 40-80% and QFR >0.8
5. Target lesion must have a visually estimated diameter of 2.0-4.0 mm and length of ≤ 50 mm
6. Target lesion must have any two of the intravascular imaging criteria of PB >65%, MLA <3.5 mm^2 (OCT) or 4.0mm^2 (IVUS), FCT <75 μm, or maximal lipid arc >180°
7. Subject must provide written informed consent before any study-related procedure

Exclusion Criteria:

1. Subject has known hypersensitivity or contraindication to any of the study drugs (including all asprin, P2Y12 inhibitors, one or more components of the study devices, including paclitaxel, etc) that cannot be adequately pre-medicated
2. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.)
3. Hypotension, shock, or need for mechanical support or intravenous vasopressors;
4. Creatinine clearance ≤30 ml/min/1.73 m^2 (as calculated by MDRD formula for estimated GFR)
5. Left ventricular ejection fraction<30% by the most recent imaging test within 30 days before procedure (echo, MRI, contrast left ventriculography or others)
6. Life expectancy <2 years for any
7. Subject is currently participating in another investigational drug or device clinical study that has not yet completed its primary endpoint
8. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
9. The target lesion is located within 10 mm of the proximal or distal of stent
10. The target lesion cannot be in the left main coronary artery
11. The target lesion is located in a bifurcation lesion (i.e., the diameter of the branch vessels is >2 mm with >50% of stenosis)
12. The target lesion is located in severe calcification or tortuosity of vessels
13. The target lesion involved in the ostium of LAD, LCX or RCA (within 3 mm of the ostium)
14. The target lesion is located within the bypass graft artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1860 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | At 24 months

SECONDARY OUTCOMES:
Target lesion failure (TLF) | At 30 days
Target lesion failure (TLF) | At 6 months
Target lesion failure (TLF) | At 12 months
Major cardiac adverse event (MACE) | At 30 days
  MACE is defined as the composite of all-cause death, recurrent myocardial infarction, revascularization, unplanned readmission for angina exacerbation or unstable angina
Major cardiac adverse event (MACE) | At 6 months
  MACE is defined as the composite of all-cause death, recurrent myocardial infarction, revascularization, unplanned readmission for angina exacerbation or unstable angina
Major cardiac adverse event (MACE) | At 12 months
  MACE is defined as the composite of all-cause death, recurrent myocardial infarction, revascularization, unplanned readmission for angina exacerbation or unstable angina
Major cardiac adverse event (MACE) | At 24 months
  MACE is defined as the composite of all-cause death, recurrent myocardial infarction, revascularization, unplanned readmission for angina exacerbation or unstable angina
All-cause death | At 30 days
  Any death will be recorded as all-cause death
All-cause death | At 6 months
  Any death will be recorded as all-cause death
All-cause death | At 12 months
  Any death will be recorded as all-cause death
All-cause death | At 24 months
  Any death will be recorded as all-cause death
Cardiac death and target lesion MI | At 30 days
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death and target lesion MI | At 6 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death and target lesion MI | At 12 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death and target lesion MI | At 24 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death | At 30 days
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death | At 6 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death | At 12 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Cardiac death | At 24 months
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Cardiac death is defined as any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), witnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment
Target lesion myocardial infarction | At 30 days
  Target lesion Myocardial Infarction (TL-MI) and non-TL-MI will be assessed
Target lesion myocardial infarction | At 6 months
  Target lesion Myocardial Infarction (TL-MI) and non-TL-MI will be assessed
Target lesion myocardial infarction | At 12 months
  Target lesion Myocardial Infarction (TL-MI) and non-TL-MI will be assessed
Target lesion myocardial infarction | At 24 months
  Target lesion Myocardial Infarction (TL-MI) and non-TL-MI will be assessed
Periprocedural myocardial infarction | At 30 days
  Periprocedural Myocardial Infarction (TL-MI) and non-Periprocedural will be assessed.
Periprocedural myocardial infarction | At 6 months
  Periprocedural Myocardial Infarction (TL-MI) and non-Periprocedural will be assessed.
Periprocedural myocardial infarction | At 12 months
  Periprocedural Myocardial Infarction (TL-MI) and non-Periprocedural will be assessed.
Periprocedural myocardial infarction | At 24 months
  Periprocedural Myocardial Infarction (TL-MI) and non-Periprocedural will be assessed.
Periprocedural and non-periprocedural myocardial infarction | At 30 days
  Periprocedural Myocardial Infarction (TL-MI) and non-periprocedural will be assessed
Periprocedural and non-periprocedural myocardial infarction | At 6 months
  Periprocedural Myocardial Infarction (TL-MI) and non-periprocedural will be assessed
Periprocedural and non-periprocedural myocardial infarction | At 12 months
  Periprocedural Myocardial Infarction (TL-MI) and non-periprocedural will be assessed
Periprocedural and non-periprocedural myocardial infarction | At 24 months
  Periprocedural Myocardial Infarction (TL-MI) and non-periprocedural will be assessed
Target vessel failure (TVF) | At 30 days
  TVF is defined as the composite of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization.
Target vessel failure (TVF) | At 6 months
  TVF is defined as the composite of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization.
Target vessel failure (TVF) | At 12 months
  TVF is defined as the composite of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization.
Target vessel failure (TVF) | At 24 months
  TVF is defined as the composite of cardiac death, target vessel myocardial infarction and ischemia-driven target vessel revascularization.
Minimal lumen area after DCB treatment | At baseline
  Post-procedure imaging examination is required
Plaque burden after DCB treatment | At baseline
  Post-procedure imaging examination is required
FCT after DCB treatment | At baseline
  Post-procedure imaging examination is required
Lipid arc after DCB treatment | At baseline
  Post-procedure imaging examination is required
FCT <75 μm after DCB treatment | At baseline
  Post-procedure imaging examination is required
PB >65% after DCB treatment | At baseline
  Post-procedure imaging examination is required
PB >70% after DCB treatment | At baseline
  Post-procedure imaging examination is required
MLA <3.5 mm^2 after DCB treatment | At baseline
  Post-procedure imaging examination is required
Maximal lipid arc >180° after DCB treatment | At baseline
  Post-procedure imaging examination is required
Cardiac biomarkers: GDF-15, interleukin-6, interleukin-1β and ceramide etc. | At baseline and one-year follow-up
  The centers with sample preservation qualifications will be asked to preserve blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (18):
- China (18):
  - Affiliated Beijing Luhe Hospital of Capital Medical University, Beijin, Beijing Municipality
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Mudanjiang Cardiovascular Hospital, Mudanjiang, Heilongjiang
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - The Third Second Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The People's Hospital of Liaoning Province, Shengyang, Liaoning
  - The Affiliated Hospital of Neimenggu Medical University, Hohhot, Neimenggu
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong